CLINICAL TRIAL: NCT03038438
Title: A Multi-center, Non-randomized Study to Evaluate the Safety and Effectiveness of the Abre Venous Self-expanding Stent System in Patients With Symptomatic Iliofemoral Venous Outflow Obstruction
Brief Title: ABRE Clinical Study of the Abre Venous Self-expanding Stent System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APV-ABRE
Record Dates: First submitted 2017-01-28; First posted 2017-01-31 (Estimated); Results first posted 2021-03-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Iliofemoral Venous Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Abre (Experimental): Abre Venous Self-expanding Stent System
  Interventions: Device: Abre venous self-expanding stent system

INTERVENTIONS:
Device: Abre venous self-expanding stent system — venous stent

SUMMARY:
Evaluate the safety and effectiveness of the Abre venous self-expanding stent system for treatment of symptomatic iliofemoral venous outflow obstruction in patients with venous occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 and ≤ 80 years of age;
2. Patient has at least one of the following clinical manifestations (i.e. symptoms and/or signs) of venous disease in lower extremity:

   * CEAP score ≥ 3
   * Venous Clinical Severity Score pain score (VCSS) ≥2
   * Suspected deep vein thrombosis (DVT);
3. Patient is willing and capable of complying with specified follow-up evaluations at the specified times;
4. Patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Ethics Board.
5. Patient has diagnosis of non-malignant venous obstruction within the common iliac, external iliac, and/or common femoral vein. The proximal point of the obstruction may extend to the iliac venous confluence of the inferior vena cava and the distal point may be at or above the deep femoral vein. Diagnosis must be made based on objective imaging by using venography and/or intravascular ultrasound (IVUS);
6. Patient has an obstructive lesion defined as:

   * Occluded, or
   * ≥50% in diameter reduction on venography or IVUS, or
   * ≥50% area reduction on IVUS
7. Acute DVT patients should be treated with the Abre stent within 14 days after onset of symptoms. Patients with acute DVT must first undergo successful treatment of acute thrombus by catheter based techniques; successful treatment is defined as 30% or less residual thrombus by venogram, as determined by physician, no bleeding, no symptomatic pulmonary embolism (confirmed by imaging), and no renal compromise (renal compromise defined as GFR>30). Patients with underlying obstructive lesions can then be included in the study within the same procedure;
8. Target vessel can accommodate a 9 French Sheath, from insertion site to target segment;
9. Exchangeable guidewire must cross target lesion(s) with successful predilation.

Exclusion Criteria:

1. Patient with DVT in the target limb of which the onset of symptoms is between 15 days and 6 months prior to planned treatment or patient has an acute DVT anywhere else than in the target vessel;
2. Patient has peripheral arterial disease causing symptoms in target limb;
3. Patient is pregnant, female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure;
4. Patient has a known or suspected systemic infection at the time of the index procedure;
5. Patient has a planned percutaneous or surgical intervention within 30 days prior or 30 days following index procedure, or a contralateral iliofemoral lesion requiring planned treatment within 12 months;
6. Patient requires femoral endovenectomy and patch venoplasty, greater saphenous vein ablation, and/or small saphenous vein stripping during the index procedure;
7. Patient has an active vasculitic inflammatory disorder (e.g. Behcet disease) predisposing the patient to thrombosis and requiring systemic corticosteroid therapy;
8. Patient has impaired renal function (GFR < 30) or is on dialysis;
9. Patient has a platelet count < 50,000 cells/mm3 or > 1,000,000 cells/mm3 and/or a White Blood Cell count < 3,000 cells/mm3 or > 12,500 cells/mm3;
10. Patient has a history of bleeding diathesis or either a history or presence of heparin induced thrombocytopenia antibodies;
11. Patient has a known hypersensitivity or contraindication to antiplatelets or anticoagulation, nitinol, or a contrast sensitivity that cannot be adequately pre-medicated;
12. Patient has presence of other severe co-morbid conditions, which in the investigator's opinion may interfere with the patient's compliance with study visits and procedures, or may confound interpretation of study data (e.g. congestive heart failure Class III and IV, non-ambulatory patients, severe hepatic dysfunction, life expectancy < 1 year);
13. Patient belongs to a vulnerable population per investigator's judgment or patient has any kind of disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures. Patient must be able to consent for themselves;
14. Patient is currently participating in another investigational drug or device study or observational competitive study.
15. Patient has a vena cava obstruction or lesion extending into the inferior vena cava (IVC), or the presence of bilateral iliofemoral venous lesions requiring planned treatment within 12 months;
16. Patient has significant venous bleeding, arterial dissection or other injury requiring additional percutaneous or surgical intervention prior to enrollment;
17. Patient has a previously placed stent in the ipsilateral venous vasculature;
18. Patient has disease that precludes safe advancement of the venous stent to the target lesion(s)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Murphy, MD, Principal Investigator — Carolinas Health Care System; Stephen Black, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (24):
- United States (16):
  - St. Joseph Hospital, Orange, California
  - The Vascular Experts, Darien, Connecticut
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Holy Name Medical Center, Teaneck, New Jersey
  - Albany Medical Center, Albany, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Health System, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - Cardiac Center of Texas, McKinney, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Lake Washington Vascular, PLLC, Bellevue, Washington
- France (2):
  - Assistance Publique - Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Hôpital Européen Georges Pompidou, Paris
- Germany (2):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Arnsberg, Karolinen Hospital, Arnsberg
- Galway University Hospitals - University Hospital Galway, Galway, Ireland
- Hesperia Hospital, Modena, Italy
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust - University College London Hospitals, London
  - Guy's & St Thomas' NHS Foundation Trust - St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy E, Gibson K, Sapoval M, Dexter DJ, Kolluri R, Razavi M, Black S. Pivotal Study Evaluating the Safety and Effectiveness of the Abre Venous Self-Expanding Stent System in Patients With Symptomatic Iliofemoral Venous Outflow Obstruction. Circ Cardiovasc Interv. 2022 Feb;15(2):e010960. doi: 10.1161/CIRCINTERVENTIONS.121.010960. Epub 2022 Feb 2. PMID 35105153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for enrollment based on the study Inclusion/Exclusion criteria between December 2017 and November 2018. Included subjects went on to have one or more Abre stents implanted. The first subject was included on December 19, 2017 and the last subject was included on November 29, 2018.
Pre-assignment Details: Of the 260 enrolled subjects, 200 met inclusion criteria and were implanted with the Abre stent(s).
Groups:
- ABRE: Subjects implanted with one or more Abre stents.
Period: Overall Study
Arm/Group | ABRE
Started | 200
30-Day Follow-Up | 198
6-Month Follow-up | 193
12-Month Follow-up | 191
24-Month Follow-up | 148
36-Month Follow-up | 162
Completed | 162
Not Completed | 38
Not completed — Death | 3
Not completed — Lost to Follow-up | 8
Not completed — Subject Incarcerated, Moved, or Refused | 4
Not completed — Withdrawal by Subject | 5
Not completed — No 36-Month Follow-Up | 18

BASELINE CHARACTERISTICS:
Groups:
- ABRE: Subjects included and implanted with one or more Abre stents
Arm/Group | ABRE
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 160
  Unknown or Not Reported | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 157
  More than one race | 0
  Unknown or Not Reported | 22
Region of Enrollment [Number; unit: participants]
  United States | 128
  Ireland | 5
  United Kingdom | 28
  Italy | 6
  France | 22
  Germany | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency
Description: Freedom from occlusion of the stented segment; Freedom from restenosis >=50%; and Freedom from clinically-driven target lesion revascularization
Time Frame: 12 Months
Population: Proportion Rate
Measure: Count of Participants; unit: Participants
Arm/Group | ABRE
Number analyzed (Participants) | 184
Participants | 162
Statistical Analysis 1: Comparison: ABRE; The primary effectiveness endpoint, primary patency at 12 months, was tested against a PG of 75%. The null and alternative hypotheses tested appear below: H0: π ≤ PG vs. HA: π > PG where π is the primary patency rate at 12 months in the study population and PG is the performance goal of 75%. The primary effectiveness objective will be met if the lower limit of the 97.5% one-sided confidence interval is above 75%; Test type: Other — Single arm study with a hypothesis test comparing to performance goal; p < 0.0001, Fisher Exact; Proportion = 88.0, 97.5% CI 1-sided [lower limit 82.5]

2. Primary Outcome: Composite Major Adverse Events
Description: The components of the Major Adverse Events include:
  All-cause death occurring post-procedure, clinically-significant pulmonary embolism, major bleeding complication, stent thrombosis, and stent migration
Time Frame: 30 Days
Population: Proportion Rate
Measure: Count of Participants; unit: Participants
Arm/Group | ABRE
Number analyzed (Participants) | 200
Participants | 4
Statistical Analysis 1: Comparison: ABRE; The primary safety endpoint, major adverse events at 30 days post-procedure, was tested against a performance goal of 12.5%. The null and alternative hypotheses tested appear below: H0: P ≥ PG vs. HA: P < PG where P is the primary safety endpoint at 30 days in the study population and PG is the performance goal. The primary safety objective will be met if the upper limit of the 97.5% one-sided confidence interval is below 12.5%; Test type: Other — Single-arm study with a hypothesis test comparing to performance goal; p < 0.0001, Fisher Exact; Proportion = 2.0, 97.5% CI 1-sided [upper limit 5.0]

3. Secondary Outcome: Device Success
Description: Successful delivery and deployment of the stent and removal of the delivery system during the index procedure. Stent based outcome measure.
Time Frame: Index Procedure
Population: 302 Abre stents were implanted in 200 included subjects.
Measure: Count of Units; unit: Implanted Stents
Units Other Than Participants: Implanted Stents
Arm/Group | ABRE
Number analyzed (Participants) | 200
Number analyzed (Implanted Stents) | 302
Implanted Stents | 302

4. Secondary Outcome: Lesion Success Obtained at Index Procedure
Description: Venographic evidence of <50% residual stenosis of the stented segment of the target lesion after post-dilation.
Time Frame: Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ABRE
Number analyzed (Participants) | 200
Participants | 200

5. Secondary Outcome: Index Procedure Success
Description: Lesion success without procedure-related MAEs prior to hospital discharge
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ABRE
Number analyzed (Participants) | 200
Participants | 198

6. Secondary Outcome: Primary Patency
Description: Primary Patency: Defined as meeting all of the following criteria:
  * Freedom from occlusion of the stented segment of the target lesion;
  * Freedom from restenosis ≥50% of the stented segment of the target lesion;
  * Freedom from clinically driven target lesion revascularization.
Time Frame: 24 Months, 36 Months
Population: SURVIVAL estimate using Kaplan-Meier method. Estimate made at 720 and 1080 days.
Measure: Number; unit: Event-Free %
Arm/Group | ABRE
Number analyzed (Participants) | 200
Event-Free %
  24 Months | 86.2
  36 Months | 81.6

7. Secondary Outcome: Primary Assisted Patency
Description: Uninterrupted patency of the stented segment of the target lesion with a secondary intervention, also known as an adjunctive treatment (e.g. balloon venoplasty, subsequent stenting, etc.)
Time Frame: 12 Months, 24 Months, 36 Months
Population: SURVIVAL estimate using Kaplan-Meier method. Estimate made at 360, 720, and 1080 days.
Measure: Number; unit: Event-Free %
Arm/Group | ABRE
Number analyzed (Participants) | 200
Event-Free %
  12 Months | 97.0
  24 Months | 90.2
  36 Months | 84.8

8. Secondary Outcome: Secondary Patency
Description: Secondary patency is defined as patency of the stented segment of the target lesion after subsequent intervention for an occlusion.
Time Frame: 12 Months, 24 Months, 36 Months
Population: SURVIVAL estimate using Kaplan-Meier method. Estimate made at 360, 720, and 1080 days.
Measure: Number; unit: Event-Free %
Arm/Group | ABRE
Number analyzed (Participants) | 200
Event-Free %
  12 Month | 99.0
  24 Months | 91.8
  36 Months | 86.3

9. Secondary Outcome: Stent Fracture
Description: X-ray for the 30-day visit was only required on the first 30 subjects. Stent Fracture within 12, 24, and 36 months included subjects who had scheduled visit-based evaluable imaging and unscheduled imaging up to day 420, 780, and 1080, respectively.
Time Frame: 30 Days, 12 Months, 24 Months, 36 Months
Population: X-ray for the 30-day visit was only required on the first 30 subjects; included subjects who had scheduled visit-based evaluable imaging and unscheduled imaging up to 420 days for 12 months assessment, up to 780 days for 24 months assessment, and up to 1140 days for 36 months assessment.
Measure: Number; unit: Stents
Units Other Than Participants: Stents
Arm/Group | ABRE
Number analyzed (Participants) | 200
Number analyzed (Stents) | 302
Stents
  30 Day: number analyzed (Participants) | 30
  30 Day: number analyzed (Stents) | 47
  30 Day | 0
  12 Months: number analyzed (Participants) | 180
  12 Months: number analyzed (Stents) | 270
  12 Months | 0
  24 Months: number analyzed (Participants) | 130
  24 Months: number analyzed (Stents) | 201
  24 Months | 0
  36 Months: number analyzed (Participants) | 143
  36 Months: number analyzed (Stents) | 215
  36 Months | 0

10. Secondary Outcome: Target Lesion Revascularization
Description: Percentage of subjects with target lesion revascularization through 30 days, 180 days, 360 days, 720, and 1080 days.
Time Frame: 30 days, 6 months, 12 months, 24 months, 36 months
Population: Cumulative incidence estimate using Kaplan-Meier method. Estimate made at 30, 180, 360, 720, and 1080 days.
Measure: Number; unit: Event %
Arm/Group | ABRE
Number analyzed (Participants) | 200
Event %
  30 Days | 3.0
  6 Months | 7.5
  12 Months | 11.1
  24 Months | 14.7
  36 Months | 16.3

11. Secondary Outcome: Delayed Stent Migration
Description: Delayed Stent Migration within 12, 24, and 36 months included subjects who had scheduled visit-based evaluable imaging and unscheduled imaging up to day 420, 780, and 1140, respectively.
Time Frame: 12 Months, 24 Months, 36 Months
Population: Included subjects who had scheduled visit-based evaluable imaging and unscheduled imaging
Measure: Number; unit: Stent number
Units Other Than Participants: Stents
Arm/Group | ABRE
Number analyzed (Participants) | 200
Number analyzed (Stents) | 302
Stent number
  12 Months: number analyzed (Participants) | 181
  12 Months: number analyzed (Stents) | 271
  12 Months | 0
  24 Months: number analyzed (Participants) | 131
  24 Months: number analyzed (Stents) | 203
  24 Months | 0
  36 Months: number analyzed (Participants) | 143
  36 Months: number analyzed (Stents) | 214
  36 Months | 0

12. Secondary Outcome: Major Adverse Events
Description: Safety endpoints (MAE, TLR, and Major Bleeding) included subjects with an event or without an event but follow-up days have reached 150 days for 6-month, 330 days for 12-month, 690 days for 24-month, and 1050 days for 36-month visit.
Time Frame: 6 Months, 12 Months, 24 Months, 36 Months
Population: Cumulative incidence estimate using Kaplan-Meier method. Estimate made at 180, 360, 720, and 1080 days.
Measure: Number; unit: Event %
Arm/Group | ABRE
Number analyzed (Participants) | 200
Event %
  Within 6 Months | 4.5
  Within 12 Months | 6.0
  Within 24 Months | 8.6
  Within 36 Months | 10.2

13. Secondary Outcome: Major Bleeding Related to Index Procedure
Description: A blood loss leading to transfusion of whole blood or red cells provided hemoglobin drop of 3 g/dL (1.86 mmol/L) or more post-index procedure is related to bleeding occurring during the index procedure.
Time Frame: 30 Days, 6 Months, 12 Months, 24 Months, 36 Months
Population: Subjects with an event or a minimum number of follow-up days per time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ABRE
Number analyzed (Participants) | 200
Participants
  30 Days | 0
  6 Months: number analyzed (Participants) | 199
  6 Months | 0
  12 Months: number analyzed (Participants) | 197
  12 Months | 0
  24 Months: number analyzed (Participants) | 192
  24 Months | 0
  36 Months: number analyzed (Participants) | 177
  36 Months | 0

14. Secondary Outcome: Re-Hospitalization
Description: Number of subjects that were re-hospitalized due to their target lesion from the Index Procedure.
Time Frame: 0-180, 181-360, 361-720, 721-1080 and 0-1080 days
Population: Subjects with an event or a minimum number of follow-up days per time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ABRE
Number analyzed (Participants) | 200
Participants
  0-6 Months | 11
  6-12 Months: number analyzed (Participants) | 199
  6-12 Months | 5
  12-24 Months: number analyzed (Participants) | 196
  12-24 Months | 6
  24-36 Months: number analyzed (Participants) | 190
  24-36 Months | 5
  0-36 Months | 20

15. Secondary Outcome: Villalta Score
Description: Villalta scores categorize the severity of post-thrombotic syndrome (PTS). Higher score indicates increasing severity of PTS. A score of greater or equal to 5 indicates PTS. PTS severity: total score of 5 to 9, mild PTS; score of 10 to 14, moderate PTS; and score of greater or equal to 15 or venous ulcer present, severe PTS.
  Change in Villalta scores were calculated as the Follow-up score minus the Baseline score (6, 12, 24, or 36 months).
  A negative change is associated with improved outcome.
Time Frame: Baseline to 6 Months, 12 Months, 24 Months, 36 Months
Population: Subjects with available data at time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABRE
Number analyzed (Participants) | 200
score on a scale
  Change from Baseline to 6 Months: number analyzed (Participants) | 189
  Change from Baseline to 6 Months | -6.5 (5.4)
  Change from Baseline to 12 Months: number analyzed (Participants) | 190
  Change from Baseline to 12 Months | -7.0 (5.6)
  Change from Baseline to 24 Months: number analyzed (Participants) | 146
  Change from Baseline to 24 Months | -6.7 (6.2)
  Change from Baseline to 36 Months: number analyzed (Participants) | 159
  Change from Baseline to 36 Months | -6.3 (5.3)

16. Secondary Outcome: Venous Clinical Severity Score (VCSS)
Description: VCSS scores range from 0=no disease to 30=severe disease. Change in VCSS score was calculated as the Follow-up score minus the Baseline score.
  A negative change is associated with improved outcome.
Time Frame: Baseline to 6 Months, 12 Months, 24 Months, 36 Months
Population: Subjects with available data at time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABRE
Number analyzed (Participants) | 200
score on a scale
  Change from Baseline to 6 Months: number analyzed (Participants) | 190
  Change from Baseline to 6 Months | -4.0 (3.7)
  Change from Baseline to 12 Months: number analyzed (Participants) | 191
  Change from Baseline to 12 Months | -4.6 (4.3)
  Change from Baseline to 24 Months: number analyzed (Participants) | 147
  Change from Baseline to 24 Months | -4.8 (4.4)
  Change from Baseline to 36 Months: number analyzed (Participants) | 160
  Change from Baseline to 36 Months | -4.5 (3.9)

17. Secondary Outcome: EuroQol-5 Dimension (EQ-5D) Score
Description: Higher score indicates a better quality of life. The questionnaire contains five dimensions where scores rank from 1 (best) to 5 (worst) plus a visual analog scale (VAS) (0 = worst health; 100 = best health).
  A positive change is associated with improved outcome. Change in EQ-5D scores were calculated as the Follow-up score minus the Baseline score (6, 12, 24, and 24 months) for both the index and VAS scores.
Time Frame: Baseline to 6 Months, 12 Months, 24 Months, 36 Months
Population: Subjects with available data at time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABRE
Number analyzed (Participants) | 200
score on a scale
  EQ-5D Index Score change from Baseline to 6 Months: number analyzed (Participants) | 192
  EQ-5D Index Score change from Baseline to 6 Months | 0.15 (0.23)
  EQ-5D Index Score change from Baseline to 12 Months: number analyzed (Participants) | 192
  EQ-5D Index Score change from Baseline to 12 Months | 0.14 (0.26)
  EQ-5D Index Score change from Baseline to 24 Months: number analyzed (Participants) | 147
  EQ-5D Index Score change from Baseline to 24 Months | 0.12 (0.26)
  EQ-5D Index Score change from Baseline to 36 Months: number analyzed (Participants) | 159
  EQ-5D Index Score change from Baseline to 36 Months | 0.13 (0.24)
  EQ-5D VAS change from baseline to 6 Months: number analyzed (Participants) | 192
  EQ-5D VAS change from baseline to 6 Months | 9.3 (22.0)
  EQ-5D VAS change from baseline to 12 Months: number analyzed (Participants) | 191
  EQ-5D VAS change from baseline to 12 Months | 8.6 (23.1)
  EQ-5D VAS change from baseline to 24 Months: number analyzed (Participants) | 146
  EQ-5D VAS change from baseline to 24 Months | 9.7 (20.3)
  EQ-5D VAS change from baseline to 36 Months: number analyzed (Participants) | 158
  EQ-5D VAS change from baseline to 36 Months | 7.7 (23.7)

18. Secondary Outcome: Venous Insufficiency Epidemiological and Economic Study (VEINES) - Quality of Life/Symptoms (QOL/Sym) Score
Description: Venous Insufficiency Epidemiological and Economic Study (VEINES) - Quality of Life/Symptoms (QOL/Sym).
  Higher scores correlate to better quality of life on a scale of 1-100. Change in VEINES QOL/Sym scores were calculated as the Follow-up score minus the Baseline score (6, 12, 24, or 36 months).
  A positive change is associated with improved outcome.
Time Frame: Change from Baseline to 6 Months, 12 Months, 24 Months, 36 Months
Population: Subjects with available data at time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABRE
Number analyzed (Participants) | 200
score on a scale
  VEINES QoL change from Baseline to 6 Months: number analyzed (Participants) | 192
  VEINES QoL change from Baseline to 6 Months | 22.2 (25.3)
  VEINES QoL change from Baseline to 12 Months: number analyzed (Participants) | 192
  VEINES QoL change from Baseline to 12 Months | 22.9 (25.1)
  VEINES QoL change from Baseline to 24 Months: number analyzed (Participants) | 148
  VEINES QoL change from Baseline to 24 Months | 21.8 (28.1)
  VEINES QoL change from Baseline to 36 Months: number analyzed (Participants) | 155
  VEINES QoL change from Baseline to 36 Months | 21.4 (25.2)
  VEINES Sym change from Baseline to 6 months: number analyzed (Participants) | 192
  VEINES Sym change from Baseline to 6 months | 22.3 (23.6)
  VEINES Sym change from Baseline to 12 months: number analyzed (Participants) | 192
  VEINES Sym change from Baseline to 12 months | 20.9 (24.0)
  VEINES Sym change from Baseline to 24 months: number analyzed (Participants) | 148
  VEINES Sym change from Baseline to 24 months | 20.4 (26.9)
  VEINES Sym change from Baseline to 36 months: number analyzed (Participants) | 155
  VEINES Sym change from Baseline to 36 months | 20.2 (24.9)

ADVERSE EVENTS:
Time Frame: Through 1080 Days
Arm/Group | ABRE
All-Cause Mortality (participants affected / at risk) | 3/200
Serious Adverse Events (participants affected / at risk) | 86/200
Other Adverse Events (participants affected / at risk) | 17/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABRE (N=200)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 5 (6)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 (3)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
BRCA2 GENE MUTATION (Congenital, familial and genetic disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 2 (2)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 1 (1)
ANAL FISSURE (Gastrointestinal disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1)
PERIPHERAL SWELLING (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
VASCULAR STENT OCCLUSION (General disorders) | 1 (1)
VASCULAR STENT STENOSIS (General disorders) | 11 (14)
VASCULAR STENT THROMBOSIS (General disorders) | 24 (35)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 7 (8)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 2 (2)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
VASCULAR ACCESS SITE HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2)
VASCULAR ACCESS SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (2)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NONKERATINISING CARCINOMA OF NASOPHARYNX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
CERVICAL RADICULOPATHY (Nervous system disorders) | 1 (1)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1)
MYELOPATHY (Nervous system disorders) | 1 (1)
VASCULAR DEMENTIA (Nervous system disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 1 (1)
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 1 (1)
UTEROVAGINAL PROLAPSE (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (2)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (3)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 4 (4)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
COLLATERAL CIRCULATION (Vascular disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 6 (15)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2)
LYMPHOEDEMA (Vascular disorders) | 2 (2)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (2)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 (3)
PERIPHERAL VEIN STENOSIS (Vascular disorders) | 1 (1)
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 4 (5)
VENA CAVA THROMBOSIS (Vascular disorders) | 1 (1)
VENOUS HAEMORRHAGE (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABRE (N=200)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT03038438/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT03038438/SAP_001.pdf